CLINICAL TRIAL: NCT03864094
Title: "Haemodynamic Stability During Induction of General Anesthesia With Propofol and Remifentanil: A Randomized, Controlled, Double-blind Study Comparing Equipotent Prophylactic Doses of Ephedrine, Phenylephrine, Norepinephrine vs Placebo."
Brief Title: Hemodynamics During Induction of General Anesthesia After Prophylactic Ephedrine, Phenylephrine or Norepinephrine.
Acronym: VH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Gunnar Helge Sjøen, Consultant in Anesthesiology, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019/374; 2019-000965-19 (EudraCT Number)
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Hemodynamic Instability; Anesthesia, General; Anesthesia, Intravenous
Keywords: Cardiac Output (CO); Systolic Blood Pressure (SBP); Systemic Vascular Resistance (SVR); Heart Rate (HR); Stroke Volume (SV); Lithium Dilutional Cardiac Output (LiDCO); Minimal Invasive Hemodynamic Monitor; Propofol; Remifentanil; Ephedrine; Phenylephrine; Norepinephrine
MeSH Terms: interventions — Ephedrine; Acetaminophen; Phenylephrine; Norepinephrine; Sodium Chloride; Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization made by a person not involved in trial in other ways. Allocation masked in sealed envelopes, stored in a locked cash box only opened by two drug preparing nurses not involved in patient care. Syringe labelled with patient identification (ID) (eg 04Vaso). Patient, Care Provider and Investigator blinded for actual concentration of drug. Allocation break after data data wash and processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ephedrine Propofol Remifentanil (Active Comparator): Prophylactic Ephedrine
  Interventions: Drug: Ephedrine; Drug: Propofol; Drug: Remifentanil
- Phenylephrine Propofol Remifentanil (Active Comparator): Prophylactic Phenylephrine
  Interventions: Drug: Phenylephrine; Drug: Propofol; Drug: Remifentanil
- Norepinephrine Propofol Remifentanil (Active Comparator): Prophylactic Norepinephrine
  Interventions: Drug: Norepinephrine; Drug: Propofol; Drug: Remifentanil
- Sodium chloride Propofol Remifentanil (Sham Comparator): NaCl Placebo
  Interventions: Drug: Sodium chloride; Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Ephedrine — 0,1 mg/kg
  Other Names: Ephedrine Sulphate Injection
  Arms: Ephedrine Propofol Remifentanil
Drug: Phenylephrine — 1 microg/kg
  Other Names: Phenylephrine Hydrocloride Injection
  Arms: Phenylephrine Propofol Remifentanil
Drug: Norepinephrine — 0,1 microg/kg
  Other Names: Noradrenalin
  Arms: Norepinephrine Propofol Remifentanil
Drug: Sodium chloride — 0,1 ml/kg
  Other Names: Sodium Chloride 0,9% injection
  Arms: Sodium chloride Propofol Remifentanil
Drug: Propofol — 2 mg/kg
  Other Names: Propolipid
Drug: Remifentanil — 1,7 microg/kg
  Other Names: Ultiva

SUMMARY:
In this trial the investigators want to examine if there is any difference in hemodynamic stability when giving equipotent prophylactic injections of ephedrine 0,1 mg/kg, phenylephrine 1 microg/kg, norepinephrine 0,1 microg/kg or sodium chloride (NaCl) 9 mg/ml during induction of general anesthesia with propofol and remifentanil.

DETAILED DESCRIPTION:
The LiDCOplus monitoring system (Lithium Dilutional Cardiac Output (LiDCO) Ltd., Cambridge, United Kingdom) is a minimally invasive monitor for measuring stroke volume (SV) using two different algorithms. The PulseCO (PulseCO ™, Cambridge, United Kingdom) is based on analyses of the the arterial pressure wave giving nominal values. The LiDCO uses lithium-dilution for calibration to give absolute values. In this trial, the investigators will use the PulseCO looking at relative changes in uncalibrated hemodynamic variables. Continual changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (CO) and systemic vascular resistance (SVR) will be measured.

Earlier studies have shown that propofol 2.5 mg/kg induction without opioid reduces CO (-15%), SV (-5 %), MAP (-33%) and SVR (-11%) and a slight reduction i HR. High-dose remifentanil anesthesia (2 microg/kg/min), in coronary patients reduced cardiac index (-25%), SV (-14%) and MAP (-39%) in a similar manner as propofol/remifentanil (propofol target 2 microg/ml and remifentanil 0.5 microg/kg/min), but systemic vascular resistance index decreased (-14%) in propofol/remifentanil combination.

Several procedures have been proposed to minimize the negative hemodynamic changes during induction. Administration of a crystalloid or a colloid did not prevent the decrease in MAP after induction of general anesthesia with propofol and fentanyl.

The hemodynamic effects in propofol-fentanyl anesthesia of preoperative ephedrine 0.07-0.15 mg/kg vs phenylephrine 1.5 microg/kg in valve surgery and concludes that ephedrine 0.07-0.1 mg/kg is safe and effective in counteracting hypotension. A dose of 0.15 mg/kg ephedrine is suggested for preventing hypotension during anesthesia induction with propofol 2.5 mg/kg and remifentanil 3 microg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18-50 years
* Gynecological procedures
* General anesthesia

Exclusion Criteria:

* Pre-existing hypertension
* Diabetes for several years
* Ischemic heart disease
* Cerebrovascular disease
* Heart valve disease
* Verified cardiac arrhythmia
* Anaemia
* Kidney or hepatic disease
* Hypersensitivity for soya, eggs or peanuts
* Pregnancy
* Poor health state
* Illicit substance use
* BMI <20 or >35 kg/m2
* SBP >150 mmHg
* HR >100 beats/min

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | First 7,5 minutes from start of induction
  Change in SBP during induction as measured by the LiDCOplus monitoring system
Heart Rate (HR) | First 7,5 minutes from start of induction
  Change in HR during induction as measured by the LiDCOplus monitoring system

SECONDARY OUTCOMES:
Stroke Volume (SV) | First 7,5 minutes from start of induction
  Change in SV during induction as measured by the LiDCOplus monitoring system
Cardiac Output (CO) | First 7,5 minutes from a start of induction
  Change in CO during induction as measured by the LiDCOplus monitoring system
Systemic Vascular Resistance (SVR) | First 7,5 minutes from start of induction
  Change in SVR during induction as measured by the LiDCOplus monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Sjøen, MD, Principal Investigator — Helse Fonna
Locations (1):
- Helse Fonna, Haugesund Sykehus, Haugesund, Norway

IPD SHARING:
Plan to Share IPD: Yes
LiDCO-csv raw data and processed data will be made public at the publishers site, and the supporting information by request to the Principal Investigator. Statistical Data Plan is included in Study Protocol.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be stored for 15 years after end of study, and may be shared during this time frame.
Access Criteria: The data may be shared by contacting the Principal Investigator.

REFERENCES:
- [Background] Fairfield JE, Dritsas A, Beale RJ. Haemodynamic effects of propofol: induction with 2.5 mg kg-1. Br J Anaesth. 1991 Nov;67(5):618-20. doi: 10.1093/bja/67.5.618. PMID 1751277
- [Background] Kazmaier S, Hanekop GG, Buhre W, Weyland A, Busch T, Radke OC, Zoelffel R, Sonntag H. Myocardial consequences of remifentanil in patients with coronary artery disease. Br J Anaesth. 2000 May;84(5):578-83. doi: 10.1093/bja/84.5.578. PMID 10844832
- [Background] Turner RJ, Gatt SP, Kam PC, Ramzan I, Daley M. Administration of a crystalloid fluid preload does not prevent the decrease in arterial blood pressure after induction of anaesthesia with propofol and fentanyl. Br J Anaesth. 1998 Jun;80(6):737-41. doi: 10.1093/bja/80.6.737. PMID 9771299
- [Background] Al-Ghamdi A. Hydroxyethylstarch 6% preload does not prevent the hypotension following induction with propofol and fentanyl. Middle East J Anaesthesiol. 2004 Jun;17(5):959-68. PMID 15449752
- [Background] El-Tahan MR. Preoperative ephedrine counters hypotension with propofol anesthesia during valve surgery: a dose dependent study. Ann Card Anaesth. 2011 Jan-Apr;14(1):30-40. doi: 10.4103/0971-9784.74397. PMID 21196672
- [Background] Masjedi M, Zand F, Kazemi AP, Hoseinipour A. Prophylactic effect of ephedrine to reduce hemodynamic changes associated with anesthesia induction with propofol and remifentanil. J Anaesthesiol Clin Pharmacol. 2014 Apr;30(2):217-21. doi: 10.4103/0970-9185.130024. PMID 24803761
- [Derived] Sjoen GH, Hauge TH, Falk RS, Tonnessen TI, Langesaeter E. Haemodynamic Changes After Prophylactic Doses of Ephedrine, Phenylephrine, Norepinephrine Versus Placebo During Induction of General Anaesthesia: A Randomised Trial. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70138. doi: 10.1111/aas.70138. PMID 41144827